CLINICAL TRIAL: NCT04904003
Title: Prosthetic Use, Mobility and Daily Functioning
Acronym: ProMob
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Sophies Minde Ortopedi (Industry); UniCare Bakke AS (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/2577
Record Dates: First submitted 2021-05-05; First posted 2021-05-27 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-06

CONDITIONS: Lower Leg Amputations
Keywords: Rehabilitation; Prosthetic mobility; Outcome measures

STUDY DESIGN:
Intervention Model Description: One explorative group, one intervention group and one control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experienced LLA - intervention (Experimental): Experienced lower-limb amputees that complete a 4-week semi-structured individualized rehabilitation regime with extensive testing before and after the intervention.
  Interventions: Other: Rehabilitation Intervention
- Experienced LLA - controls (Experimental): Experienced lower-limb amputees that will be tested with a 4-week interval. No intervention. This group will be matched to the group of experienced lower-limb amputees.
  Interventions: Other: Rehabilitation Intervention
- New LLA learning to use prosthesis (Experimental): New lower-limb amputees that complete a 8-11 weeks semi-structured individualized rehabilitation regime with extensive testing before and after the intervention.
  Interventions: Other: Rehabilitation Intervention

INTERVENTIONS:
Other: Rehabilitation Intervention — Strength, flexibility, endurance, balance, mobility, (self-efficacy)

SUMMARY:
The goal of the project is to explore which elements of rehabilitation that influence mobility in new and experienced unilateral lower-limb amputees.

DETAILED DESCRIPTION:
Both new and experienced unilateral lower limb amputees (LLA) describe difficulties when ambulating intentionally and independently from one place to another using prosthesis. In LLA, this decreased ability to mobilize affect daily functioning and may result in low activity-levels, impeded social participation and reduced health-related quality of life.

Both primary and secondary rehabilitation of LLA have implications for functional mobility. The consensus among health professionals is that LLA should train to improve their ability to ambulate. However, knowledge from research regarding which elements that constitute effective training and how systematic exercise affects body structures, functions, activity and participation in lower limb amputees, is limited.

There also is a lack of knowledge of how prosthetic users endure and process the challenges regarding mobility, how they adapt to the use of their prosthesis, how safe they are ambulating using the prosthesis, and how pain and psychosocial issues affect their perceived health and mobility.

The aim of this Ph.D.-project is to explore how a period of semi-standardized individualized rehabilitation originating from an evidence-based approach, affect the functional mobility of both new and experienced LLA, and how LLA process the loss of a limb and challenges during ambulation.

ELIGIBILITY:
Inclusion criteria for experienced users of prosthesis - intervention group:

* Unilaterally amputated (above the ankle joint / under the hip joint)
* Minimum 12 months since amputation
* Have a well-adapted prosthesis before baseline measurements
* Not attended an organized, regular training program for the last 6 months
* Uses the prosthesis on a daily basis
* Participation approved by physician

Inclusion Criteria for experienced users of prosthesis - control group:

* Unilaterally amputated (above the ankle joint / under the hip joint)
* Minimum 12 months since amputation
* Have a well-adapted prosthesis before baseline measurements
* Daily use of the prosthesis
* Not attended an organized, regular training program in the last 6 months
* No participation in regular and systematic training between pre- and post-testing

Inclusion Criteria for new users of prosthesis:

* Unilaterally amputated (above the ankle joint / under the hip joint)
* No prior record of use of prosthesis
* Participation approved by physician

Exclusion Criteria:

* Bilaterally amputated over ankle joint
* Lack of understanding of Norwegian language (oral, written)
* Neurological disorders affecting gait function
* Skin lesion or abrasion on the stump or remaining extremity affecting mobility and function
* Other issues that complicate participation in a rehabilitation intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Prosthetic Limb Users Survey of Mobility (Plus-M) Short form - 12 items | 4-8 weeks
  A questionnaire that measures different aspects of mobility in lower-limb amputees (LLA) using prosthesis. PLUS-M provide a score range from 17.5 to 76.6. High scores indicate better outcome.
The Amputee Mobility Predictor (AMP). | 4-8 weeks
  The test is designed to measure mobility and ability to move with prosthesis (AMPPro) and without prosthesis (AMPNoPro). AMPPro provide a score range from 0-47. AMPNoPro provide a score range from 0-43. High scores indicate better outcome.

OTHER OUTCOMES:
Trinity Amputation and Prosthesis Experience Scale-Revised (TAPES-R) - psychosocial adjustment | 4-8 weeks
  The questionnaire examines psychosocial processes involved in adapting to the prosthesis as well as specific needs when using prosthesis.
  Psychosocial adjustment - general subscale, provide a score range from 1.0-4.0. High scores indicative of positive adjustment.
  Psychosocial adjustment - social subscale, provide a score range from 1.0-4.0. High scores indicative of positive adjustment.
  Psychosocial adjustment - adjustment to limitation subscale, provide a score range from 1.0-4.0. High scores indicative of positive adjustment.
Trinity Amputation and Prosthesis Experience Scale-Revised (TAPES-R) - activity restriction scale | 4-8 weeks
  The questionnaire examines psychosocial processes involved in adapting to the prosthesis as well as specific needs when using prosthesis.
  Activity restriction scale, provide a score range from 0.0-2.0. High scores is indicative of activity restriction.
Trinity Amputation and Prosthesis Experience Scale-Revised (TAPES-R) - satisfaction with prosthesis | 4-8 weeks
  The questionnaire examines psychosocial processes involved in adapting to the prosthesis as well as specific needs when using prosthesis.
  Satisfaction with prosthesis - aesthetic satisfaction subscale, provide a score range from 3-9. High scores is indicative of satisfaction with prosthesis.
  Satisfaction with prosthesis - functional satisfaction subscale, provide a score range from 5-15. High scores is indicative of satisfaction with prosthesis.
Activities-Specific Balance Confidence scale (ABC) | 4-8 weeks
  The questionnaire measures how confident LLA are in performing ADL without losing balance or becoming unsteady. ABC provide a score range from 0-64. High scores indicate better outcome.
EuroQoL 5L - health-related quality of life (EQ-5D-5L) | 4-8 weeks
  Standardized generic instrument used to measure health outcomes and health-related quality of life. Each question provide a score range from 1-5. High scores indicate worse outcome.
Two-minute walk test (2WT) | 4-8 weeks
  The test measures functional mobility and the distance covered in two minutes.
The L-Test of Functional Mobility (L-test) | 4-8 weeks
  The test measures functional mobility and is designed specifically for LLA. The LLA walks as fast as possible in a 3 x 7 meter L-shaped walkway that requires change of direction both ways.
General Perceived Self-Efficacy Scale (GSE) | 4-8 weeks
  Assesses self-efficacy when coping with challenging demands in life. GSE provide a score range from 10-40. High scores indicate better outcome.
Grip strength | 4-8 weeks
  Grip strength as measured by hand dynamometer
Balance | 4-8 weeks
  Postural balance measured as center of pressure excursion by insoles with pressure sensors and a gyroscope sensor.
Activity level | 4-8 weeks
  Number of steps measured by an accelerometer
Gait characteristics - temporal parameters | 4-8 weeks
  Gait characteristics measured in seconds by insoles with pressure sensors and gyroscope sensor
Gait characteristics - spatial parameters | 4-8 weeks
  Gait characteristics measured in meters by insoles with pressure sensors and gyroscope sensor
Gait characteristics - ground reaction force Gait characteristics - ground reaction force | 4-8 weeks
  Gait characteristics measured in Newton by insoles with pressure sensors and gyroscope sensor

CONTACTS AND LOCATIONS:
Overall Officials: Terje Gjøvaag, PhD., Study Director — Associate professor and Head of research group
Locations (2):
- Norway (2):
  - Unicare Bakke, Halden, Akershus
  - OsloMet, Oslo

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available. The GDPR-regulations make sharing of research data both time-consuming and difficult.